CLINICAL TRIAL: NCT02985385
Title: Palliative Therapy For Lethal Congenital Malformations: An Islamic Perspective
Brief Title: Lethal Congenital Malformations: Palliative Therapy From An Islamic Point of View
Acronym: LCM
Status: Completed | Type: Observational
Sponsor: Security Forces Hospital (Other)
Responsible Party: Principal Investigator, OMER B ABDELBASIT, Principal Investigator, Security Forces Hospital
Other Study IDs: SFH
Record Dates: First submitted 2016-11-17; First posted 2016-12-07 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Congenital Malformations
Keywords: Congenital Lethal Malformations
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Abnormal Fetal Ultrasounds: Abnormal fetal ultrasounds:
  1. Those consistent with lethal malformations are provided with palliative management without providing respiratory support. Are given feeding and oxygen
  2. Those compatible with life are managed by full investigation and given standard care for each case
  Interventions: Other: Palliative management
- Normal Fetal Ultrasounds: Given normal care

INTERVENTIONS:
Other: Palliative management — Diagnostic studies for abnormal fetal ultrasounds
  Groups: Abnormal Fetal Ultrasounds

SUMMARY:
To prove that palliative therapy can be practised for congenital lethal malformations within the Islamic Code of Ethics.

After defining lethal malformation no respiratory support is offered and newborns are provided with compassionate care.

DETAILED DESCRIPTION:
This is a prospective observational study where all abnormal antenatal ultrasounds are discussed in a weekly prenatal meeting and plans are drawn for management of these abnormal fetal findings. Lethal malformations are defined as conditions which will end in death regardless of supportive care. Cases are discussed extensively and parents are involved in management decisions. When a decision of non- intervention is reached for a lethal malformation consent of the family is obtained and a plan of non monitoring for the mother is documented together with no resuscitation for the newborn. Families who do not consent to such plan are offered full support for the pregnant mother and her newborn. A record of all cases is kept available together with the management plan so that the appropriate action is taken when the the pregnant lady presents for admission. All babies with lethal malformations are recorded whether stillborn or live born and their diagnosis is confirmed. Survival time is recorded for each case.

ELIGIBILITY:
Inclusion Criteria:All babies with abnormal fetal ultrasounds -

Exclusion Criteria: Normal babies who die in the neonatal period because of other causes not associated with lethal malformations

-

Ages: 1 Hour to 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Babies with abnormal fetal ultrasounds and who fall into the definition of lethal congenital malformation according to the groups in our study
Sampling Method: Probability Sample
Enrollment: 25958 (Actual)
Dates: Start 2001-06; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Effective Palliative therapy in lethal malformations | Time of death in days for a baby with lethal malformation
  Provide palliative care only to those babies born with lethal congenital malformations in the form of oxygen and feeding

SECONDARY OUTCOMES:
Survival of babies with lethal malformations | Time of survival in hours or days
  Record of the time of survival for each group of lethal malformations

CONTACTS AND LOCATIONS:
Overall Officials: KHALID A ALHUUSEIN, CABP, Study Chair — Security Forces Hospital
Locations (1):
- Security Forces Hospital, Riyadh, Central, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All the results of lethal malformations are discussed with participants and the management planned approved. The outcome is explained in terms of mortality and length of survival. The feasibility of applying palliative therapy to lethal congenital malformations will enable muslim doctors to take the decision to withhold respiratory support to these cases.
  The results of the study have been sent to the Muslim Scholarly Council to review and evaluate them in relation to Islamic guidelines and hence share on the decision of withholding treatment for terminally sick patients. This will add weight to our decision to apply palliative therapy to babies with lethal congenital malformations.

REFERENCES:
- [Background] Wilkinson DJ, Thiele P, Watkins A, De Crespigny L. Fatally flawed? A review and ethical analysis of lethal congenital malformations. BJOG. 2012 Oct;119(11):1302-8. doi: 10.1111/j.1471-0528.2012.03450.x. Epub 2012 Jul 25. PMID 22827258
- [Background] El-Hazmi MA. Islamic teachings of bioethics in relation to the practice of medical genetics. Saudi Med J. 2007 Dec;28(12):1781-7. No abstract available. PMID 18060202
- [Background] Al-Aqeel AI. Ethical guidelines in genetics and genomics. An Islamic perspective. Saudi Med J. 2005 Dec;26(12):1862-70. PMID 16380763
- [Background] Islamic Figh Council of Moslim World League. Website: www.themwl.org/resolutions and recommendations of the council of the Islamic Figh Academy
- [Background] Schenker JG. Codes of perinatal ethics: an international perspective. Clin Perinatol. 2003 Mar;30(1):45-65. doi: 10.1016/s0095-5108(02)00081-7. PMID 12696785
- [Background] de Crespigny L. Words matter: nomenclature and communication in perinatal medicine. Clin Perinatol. 2003 Mar;30(1):17-25. doi: 10.1016/s0095-5108(02)00088-x. PMID 12696783
- [Background] Strong C. Fetal anomalies: ethical and legal considerations in screening, detection, and management. Clin Perinatol. 2003 Mar;30(1):113-26. doi: 10.1016/s0095-5108(02)00083-0. PMID 12696790
- [Background] Leuthner SR. Fetal palliative care. Clin Perinatol. 2004 Sep;31(3):649-65. doi: 10.1016/j.clp.2004.04.018. PMID 15325543